CLINICAL TRIAL: NCT00157482
Title: A Randomized, Prospective, Double-Blind Study to Evaluate the Effects on Lipid Profile of Combined Ezetimibe and Simvastatin Therapy as Compared to Simvastatin Alone in People With Type 2 Diabetes
Brief Title: Ezetimibe and Simvastatin in Dyslipidemia of Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mario Negri Institute for Pharmacological Research (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: ESD
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2007-02-13 (Estimated); Status verified 2006-12

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Ezetimibe; Simvastatin

INTERVENTIONS:
Drug: Ezetimibe
Drug: Simvastatin

SUMMARY:
Diabetes mellitus is becoming a global epidemic burden. Its chronic cardiovascular complications, myocardial infarction and stroke, are the main causes of death in diabetic patients. It was found that low density lipoprotein (LDL) cholesterol concentration is related to the increased coronary disease risk that could be successfully reduced by cholesterol-lowering therapy. Furthermore, preliminary evidence suggests that ameliorating dyslipidemia may be renoprotective in diabetic patients with proteinuria.

Ezetimibe is the first selective inhibitor of cholesterol absorption and it has demonstrated a high efficacy in lowering cholesterol concentration and an excellent safety profile. Preliminary data suggest that ezetimibe, combined with a drug that blocks the cholesterol synthesis (statins), could be even more effective in decreasing cholesterol concentration. The aim of this study is to evaluate whether ezetimibe-simvastatin combined therapy is superior to simvastatin monotherapy in ameliorating the lipid profile and albuminuria in type 2 diabetic patients.

DETAILED DESCRIPTION:
INTRODUCTION

Diabetes mellitus contributes substantially to the global burden of disease, with an estimated 150 million people affected worldwide and its prevalence is expected to double by 2025. Myocardial infarction and stroke are common causes of major morbidity in people with diabetes, most of whose deaths are attributed to cardiovascular causes. Recent findings provide definitive evidences that cholesterol-lowering therapy can produce substantial reductions in the risk of heart attacks, stroke and revascularizations in diabetic patients even if they do not have high blood cholesterol concentrations.

Also preliminary evidence is available that ameliorating dyslipidemia may be renoprotective in diabetic patients with proteinuria.

Ezetimibe is the first member of a class of highly selective cholesterol absorption inhibitors that effectively and potently prevents the absorption of cholesterol by inhibiting the passage of biliary and dietary cholesterol across the wall of the small intestine, without affecting absorption of other fat-soluble nutrients.

Many pre-clinical models have demonstrated the lipid-lowering and anti-atherosclerotic properties of ezetimibe as a single agent, and showed its synergistic effect in combination with HMGCoA reductase inhibitors (statins).

Phase I/II studies on patients with hypercholesterolemia have explored the safety and efficacy of ezetimibe monotherapy and co-administration with simvastatin. In these studies, combined therapy was safely and invariably more effective than single therapy in ameliorating the lipid profile.

Ezetimibe had an excellent safety profile in standard toxicity studies in pre-clinical models. Clinical studies in patients with primary hyperlipidemia have also indicated that monotherapy with ezetimibe and coadministration with a statin were both well tolerated. Whether ezetimibe-simvastatin combined therapy more effectively than simvastatin monotherapy ameliorates the lipid profile and albuminuria in people with diabetes is worth investigating. Evidence of a superior efficacy of ezetimibe-simvastatin would provide the rationale for a prospective trial aimed to explore the possibility of a superior cardioprotective and renoprotective effect of the combined therapy.

AIM

Primary:

* To compare the effect of ezetimibe-simvastatin combination (10-40mg/day) and simvastatin (40mg/day) alone on LDL-cholesterol concentrations in type 2 diabetic patients with basal total cholesterol >135mg/dl and/or concomitant lipid lowering therapy with HMGCoA reductase inhibitors.

Secondary:

* To compare the effect of the above treatments on total cholesterol, apolipoprotein A1 and B, lipoprotein (a) and triglyceride concentrations.
* To evaluate the safety profile of these two treatments.

Explorative:

To explore the hypothesis that ameliorating dyslipidemia therapy may also result in a reduction of urinary albumin excretion rate.

DESIGN

This will be a randomized, prospective, double-blind, parallel group study. Following a 4-week wash-out period from previous lipid-lowering therapy (if any) with HMGCoA reductase inhibitors or any other kinds of lipid-lowering drugs, patients will enter a two-month run-in phase with simvastatin 40mg per day. At completion of the run-in period, patients will be randomly allocated into two double-blind treatment arms, ezetimibe 10mg + simvastatin 40mg per day or placebo + simvastatin 40mg per day for a two-month treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes mellitus with stable antidiabetic treatment since at least three months
* Total cholesterol concentrations >135mg/dl and/or concomitant lipid lowering therapy with HMGCoA inhibitors
* Serum creatinine ≤1.5mg/dl
* Urinary albumin excretion rate < 200μg/min
* Written informed consent

Exclusion Criteria:

* History of myocardial infarction, stroke or hospital admission for angina within the previous 6 months
* History of percutaneous transluminal coronary angioplasty or coronary artery bypass grafting
* Clinically manifest heart failure (grade III or above according to New York Heart Association criteria)
* Poor glycemic control (HbA1C >11%)
* Primary hyperlipidemia
* Uncontrolled thyroid diseases
* Infectious disease within 4 weeks of starting
* Acute liver disease or hepatic dysfunction
* Inflammatory muscle disease or evidence of muscle problems
* Concurrent treatment with systemic steroids, androgens, cyclosporin and other immunosuppressive drugs, fibrates, high-dose niacin or cholestyramine
* Pregnancy or lactating
* Women of childbearing potential without following a scientifically accepted form of contraception
* Life-threatening conditions or terminal concomitant diseases other than diabetes
* Specific contraindications or history of hypersensitivity to the study drugs or other statins
* Legal incapacity and/or other circumstances rendering the patient unable to understand the nature, scope and possible consequence of the trial
* Evidence of an uncooperative attitude
* Any evidence that patient will not be able to complete the trial follow-up

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108
Dates: Start 2005-01; Study Completion 2006-12

PRIMARY OUTCOMES:
LDL-cholesterol, at 16 weeks of treatment. LDL-cholesterol is measured at -4, 0, 8, 12 and 16 weeks.

SECONDARY OUTCOMES:
Total cholesterol, apolipoprotein A1 and B, lipoprotein and triglycerides, at -4, 0, 8, 12 and 16 weeks
Explorative
Urinary albumin excretion, at -4, 0, 8 and 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Piero Ruggenenti, MD, Principal Investigator — Mario Negri Institute
Locations (4):
- Italy (4):
  - Hospital "Ospedali Riuniti di Bergamo" - Diabetologic Unit, Bergamo, Bergamo
  - ASl of Ponte San Pietro - Diabetologic Unit, Ponte San Pietro, Bergamo
  - Clinical Research Center for Rare Diseases, Ranica, Bergamo
  - Hospital "Treviglio Caravaggio " - Diabetologic Unit, Treviglio, Bergamo

REFERENCES:
- [Derived] Ruggenenti P, Cattaneo D, Rota S, Iliev I, Parvanova A, Diadei O, Ene-Iordache B, Ferrari S, Bossi AC, Trevisan R, Belviso A, Remuzzi G; Ezetimibe and Simvastatin in Dyslipidemia of Diabetes (ESD) Study Group. Effects of combined ezetimibe and simvastatin therapy as compared with simvastatin alone in patients with type 2 diabetes: a prospective randomized double-blind clinical trial. Diabetes Care. 2010 Sep;33(9):1954-6. doi: 10.2337/dc10-0320. Epub 2010 Jun 21. PMID 20566677